CLINICAL TRIAL: NCT00796029
Title: Plasma Concentrations, Metabolism and Excretion of 14C-paliperidone After a Single Oral Dose in Healthy Male Subjects
Brief Title: A Study of Plasma Concentrations, Metabolism and Excretion of 14C-paliperidone After a Single Oral Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004276
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mood disorders; Antipsychotic drugs: 14C-paliperidone
MeSH Terms: conditions — Schizophrenia; Mood Disorders

INTERVENTIONS:
Drug: 14C-paliperidone

SUMMARY:
The purposes of this study are to investigate the metabolic pathways of paliperidone and excretion of paliperidone and its metabolites in healthy adult male volunteers, both CYP2D6 poor and extensive metabolizers, after administration of a single 1-mg oral dose of 14C-paliperidone, to evaluate the safety and tolerability of paliperidone, and to determine the relationship between genotypes (CYP2D6, CYP3A4, CYP3A5, UGT1A1, and UGT1A6) and exposure to paliperidone and its metabolites.

DETAILED DESCRIPTION:
This study is designed as a single-center, single-dose, open-label study of the absorption, metabolism, and excretion of paliperidone in healthy men (3 extensive and 3 poor metabolizers based on CYP2D6 phenotype). Eligible volunteers will be admitted to the study center the evening before study drug administration and will remain at the study center until 168 hours after dosing (or longer if required up to a maximum of 14 days). Each volunteer will receive a single oral dose of 14C-paliperidone with total radioactivity below 1000 µSv (16 mCi). Blood samples for plasma pharmacokinetic profile will be obtained immediately before study drug administration and 0.5, 1, 1.5, 3, 6, 12, 16, 36, 48, 72, 96, 120, 144 and 168 hours postdose. Blood samples will be obtained 2, 4, 8 and 24 hours postdose for determination of 14C in whole blood. Samples for determination of serum creatinine will be obtained 2, 4, 8 and 24 hours postdose. Urine will be collected immediately prior to drug administration and from 0-4, 4-8, 8-12, 12-16, 16-24, 24-36, 36-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours after study drug administration. Fecal samples will be collected per each stool, once before study drug administration and in the period from 0-168 hours after study drug administration. Collections of urine and feces (per 24 hours) will continue beyond 168 hours, to a maximum of 336 hours (Day 15) for patients who excrete radioactivity slowly (2 latest 24-hour urine collections each greater than or equal to 2% of total radioactive dose) or have <7 feces stool samples over the 0 to 168-hour period. 14C radioactivity will be measured in plasma, urine, and feces. Aliquots of the 0- through 24 hour urine collections will be analyzed for creatinine. Plasma concentrations of paliperidone and risperidone will be determined by means of a validated LC MS/MS method. The 14C-labeled moiety in plasma and urine will be determined by liquid scintillation counting. For all plasma samples, the lower limits of quantification for paliperidone and risperidone will be 0.100 ng/mL. For all plasma and urine samples the lower limits of quantification for 14C-paliperidone will be 72 dpm/mL (=2.0n g eq/mL). The rationale for the present study with a single-dose administration of 1 mg 14C-paliperidone to healthy white men is to determine the routes of excretion for paliperidone and to elucidate the metabolic pathways and structures of predominant paliperidone metabolites. As such, this study will result in a more complete understanding of the pharmacokinetics of paliperidone in humans. Safety and tolerability will be monitored. Volunteers will receive a single oral 1 mg dose of 14C-paliperidone as a solution with a specific activity of 592 kBq/mg, resulting in an administered radioactivity of 592 kBq (or 16 µCi). The total radioactive load for the subject will remain lower than 1000 µSv.

ELIGIBILITY:
Inclusion Criteria:

* Dextromethorphan metabolic ratio of >0.345 (poor metabolizer) or <0.0255 (extensive metabolizer)
* Body Mass Index: (weight [kg]/height [m]2) between 20 and 28 kg/m2, inclusive
* Volunteers must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* Healthy based on a prestudy physical examination, medical history, ECG, the results of hematology and serum chemistry tests, and a urinalysis carried out within the 3 weeks prior to administration of study drug. If the results of the hematology tests, serum chemistry tests (except for liver enzymes and serum creatinine), or the urinalysis are not within the laboratory's reference ranges, the volunteer can be included only on the condition that the investigator judges that the deviations are not clinically significant.

Exclusion Criteria:

* Relevant history of cardiac arrhythmias, bronchospastic or cardiovascular disease (e.g., history of ischemic heart disease or cerebrovascular accident)
* respiratory, neuropsychiatric, renal, hepatic, gastrointestinal (including surgeries, and malabsorption problems), endocrine (including diabetes mellitus and thyrotoxicosis), or immunologic diseases
* parkinsonism
* or drug allergy
* History of any cancer, with the exception of basal cell carcinoma
* Have received an experimental drug or used an experimental medical device within 30 days before the planned start of treatment
* History of smoking or use of nicotine-containing substances within the last 2 months, as determined by medical history and/or volunteer's verbal report
* History of alcohol or substance abuse. Positive test results for urine drug screen or alcohol breath test upon admission to the study center on Day 1
* Positive results for any of the serology tests (hepatitis B surface antigen, human immunodeficiency virus [HIV] antibody, and hepatitis C viral antibody)
* Liver function tests or serum creatinine exceeding normal limits at screening

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2003-07; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
To investigate the metabolic pathways of paliperidone and excretion of paliperidone and its metabolites in healthy adult male volunteers,both poor and extensive metabolizers for CYP2D6,after administration of a single 1 mg oral dose of 14C paliperidone

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of paliperidone, as well as the relationship between genotypes (CYP2D6, CYP3A4, CYP3A5, UGT1A1, and UGT1A6) and exposure to paliperidone and its metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Vermeir M, Naessens I, Remmerie B, Mannens G, Hendrickx J, Sterkens P, Talluri K, Boom S, Eerdekens M, van Osselaer N, Cleton A. Absorption, metabolism, and excretion of paliperidone, a new monoaminergic antagonist, in humans. Drug Metab Dispos. 2008 Apr;36(4):769-79. doi: 10.1124/dmd.107.018275. Epub 2008 Jan 28. PMID 18227146
- See also: A study of plasma concentrations, metabolism and excretion of 14C-paliperidone after a single oral dose — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=577&filename=CR004276_CSR.pdf